CLINICAL TRIAL: NCT02898259
Title: A Phase IB/II Trial of Lenalidomide (Revlimid®), Ixazomib and Rituximab (RIXAR) as Front-line Therapy for High Risk Indolent B Cell Lymphoma
Brief Title: Lenalidomide, Ixazomib, and Rituximab as Front-Line Therapy for High Risk Indolent B-Cell Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding was eliminated.
Sponsor: Brian Hill (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Brian Hill, MD,PhD, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1414
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Results first posted 2021-01-13 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: B Cell Lymphoma; Lymphoma
Keywords: Lenalidomide; Ixazomib; Rituximab
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma | interventions — ixazomib; Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenalidomide + Ixazomib + Rituximab (Experimental): Ixazomib will be orally administered with a starting dose of 2.0mg. Lenalidomide will be administered orally with a starting dose of 20mg. Rituximab will be administered intravenously at the standard dose of 375mg/m2. The study will use a standard 3 + 3 design for determination of MTD during cycle 1. There will be three dose levels for escalation, followed by two expansion cohorts of 12 patients each at the MTD, one cohort with follicular lymphoma and one cohort with non-follicular low-grade lymphoma (SLL, marginal zone, lymphoplasmacytic). Patients will be treated for 12 cycles of 4 week duration.
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Ixazomib — The prescribed administration of ixazomib doses in this study is 2.0, 3.0 or 4.0 mg ixazomib on days 1, 8 and 15 of each 28 day cycle.
Drug: Lenalidomide — Lenalidomide starting dose will be based on baseline calculated creatinine clearance as follows:
  * Starting lenalidomide Dose (20mg)
  * Calculated Creatinine Clearance: >=60ml/min receive 20 mg daily on Days 1 - 21 of each 28-day cycle
  * Calculated Creatinine Clearance: >= 30 and < 60 ml/min receive 10 mg daily on Days 1 - 21 of each 28-day cycle
  Other Names: Revlimid
Drug: Rituximab — Rituximab is administered intravenously at 375mg/m2 on days 1, 8, and 15 of cycle 1, day 1 of cycles 2-6 and day 1 of cycles 8, 10, and 12.
  Other Names: Rituxan

SUMMARY:
A Phase IB/II Trial of Lenalidomide (Revlimid®), Ixazomib and Rituximab (RIXAR) as Front-line Therapy for High Risk Indolent B cell Lymphoma

DETAILED DESCRIPTION:
Primary:

To determine the maximum tolerated dose and toxicity of the combination of oral ixazomib and lenalidomide plus rituximab in patients with previously untreated low-grade B cell lymphoma having high tumor burden by GELF criteria or FLIPI 3-5

Secondary:

* To determine overall response rate in an expanded cohort at the MTD for follicular lymphoma and for non-follicular low-grade B cell lymphoma
* Duration of response, time to progression, progression free survival, time to treatment failure and overall survival
* Create tissue microarray from paraffin embedded tissue for future studies.
* Assessment of baseline lymphocyte subsets as prognostic markers.

Overview of Study Design:

This study combines three classes of agents that have non-overlapping mechanisms of action and toxicity profiles, with each pair having demonstrated clinical evidence of benefit without unexpected toxicity. We use the lenalidomide-rituximab backbone, feasible and active in lymphoma, and add a novel oral proteasome inhibitor to potentially enhance efficacy, minimize toxicity and limit patient visits for treatment.

Patients with previously untreated low-grade B cell lymphoma having high tumor burden by GELF criteria or FLIPI 3-5 will be treated with the combination of oral ixazomib + lenalidomide + rituximab.

The primary objective is to determine the maximum tolerated dose and toxicity of this regimen. The study will use a standard 3 + 3 design for determination of MTD during cycle 1. There will be three dose levels for escalation, followed by two expansion cohorts of 12 patients each at the MTD, one cohort with follicular lymphoma and one cohort with non-follicular low-grade lymphoma (SLL, marginal zone, lymphoplasmacytic).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed, low-grade B-lymphocyte Non-Hodgkin's Lymphoma (NHL) by the World Health Organization Classification:

  * Follicular lymphoma grades 1, 2, and 3a
  * Marginal zone B-cell lymphoma, including extranodal (MALT), nodal and splenic. Excluding: Small lymphocytic lymphoma Lymphoplasmacytic lymphoma/Waldenström's macroglobulinemia (WM)
  * Lymphoplasmacytic lymphoma (including Waldenström's macroglobulinemia (WM))
* Must have stage 2, 3 or 4 disease, with either high tumor burden by Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria and/or Follicular Lymphoma International Prognostic Index (FLIPI) 3-5

  * To meet GELF criteria, patient must have at least one criterion:

    * Nodal or extranodal mass > 7 cm
    * At least 3 nodal masses: each > 3.0 cm in longest dimension
    * Systemic symptoms due to lymphoma or B symptoms
    * Splenomegaly with spleen > 16 cm by Computed Tomography (CT) scan
    * Evidence of compression syndrome (e.g., ureteral, orbital, gastrointestinal) or pleural or peritoneal serous effusion due to lymphoma (irrespective of cell content)
    * Leukemic presentation (> 5.0 x 10^9/L malignant circulating follicular or lymphoma cells)
    * Cytopenias (absolute neutrophil count < 1.0 X 10^9/L, hemoglobin < 10 gm/dL, and/or platelets <100 x 10^9/L).
  * AND/OR To meet FLIPI criteria, patient must have at least 3 out of the following 5 criteria:

    * Age > 60 years
    * Ann Arbor stage III-IV
    * Hemoglobin level < 12 mg/dL
    * ≥ 5 nodal areas
    * Serum Lactate Dehydrogenase (LDH) level above normal
* Must have previously untreated lymphoma. A short (< 2 week) course of steroids for symptom palliation is permitted. Prior involved field radiotherapy for symptom palliation is permitted as long as there is measurable disease outside the radiation port. If radiotherapy has been given, there should be at least 7 days between last treatment and beginning of protocol therapy.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Patients must have adequate hematologic, hepatic, and renal function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1,000/mcL
  * Platelet count ≥ 75,000/mcL
  * Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN)
  * Aspartate Aminotransferase (AST) (SGOT) ≤ 3 x institutional upper limit of normal
  * Alanine Aminotransferase (ALT) (SGPT) ≤ 3 x institutional upper limit of normal
  * Calculated creatinine clearance ≥ 30 mL/min/1.73 m^2
* Participants must agree to ongoing anticoagulation as prophylaxis against deep vein thrombosis (DVT) using aspirin (81 or 325 mg) daily, warfarin or low molecular weight heparin, or a patient already taking another oral anticoagulant (e.g. direct thrombin inhibitors for atrial fibrillation) may continue that agent.
* All study participants must be willing to register with the mandatory RevAssist program and be willing to comply with its requirements.
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
* A woman of childbearing potential must agree to practice:

  * 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * True abstinence when this is in line with the preferred and usual lifestyle of the subject.
  * A woman of childbearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to and again within 24 hours of starting therapy with Revlimid®. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document and HIPAA consent document. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

* Patients who are receiving any other investigational agents.
* Female patients who are lactating or have a positive serum pregnancy test during the screening period.
* Major surgery within 14 days before enrollment.
* Radiotherapy within 14 days before enrollment. If the involved field is small (single nodal area), 7 days will be considered a sufficient interval between treatment and beginning of protocol therapy.
* Known central nervous system involvement.
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Systemic treatment, within 14 days before the beginning of protocol therapy, with CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent. Specifically, prior desquamating rash or erythema nodosum during prior thalidomide or other similar agents.
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib or lenalidomide including difficulty swallowing.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Patient has ≥ Grade 2 peripheral neuropathy on clinical examination during the screening period.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.
* Any prior use of Revlimid® or Velcade®.
* Known seropositivity for, or active viral infection with, Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) (unless due to vaccination), or Hepatitis C Virus (HCV). HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with lenalidomide and ixazomib. In addition, these patients are at increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Pregnant or breastfeeding women are excluded from this study because lenalidomide has known teratogenic effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with lenalidomide, breastfeeding should be discontinued if the mother is treated with lenalidomide. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2022-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hill, MD, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- DL1 (Ixazomib 2.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2); DL2 (Ixazomib 3.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2); DL3/MTD (Ixazomib 4.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2); Expansion Cohort 2: Non-Follicular Lymphoma at MTD: Ixazomib will be orally administered with a starting dose of 2.0mg. Lenalidomide will be administered orally with a starting dose of 20mg. Rituximab will be administered intravenously at the standard dose of 375mg/m2. The study will use a standard 3 + 3 design for determination of MTD during cycle 1. There will be three dose levels for escalation, followed by two expansion cohorts of 12 patients each at the MTD, one cohort with follicular lymphoma and one cohort with non-follicular low-grade lymphoma (SLL, marginal zone, lymphoplasmacytic). Patients will be treated for 12 cycles of 4 week duration.
- Expansion Cohort I: Follicular Lymphoma at MTD: Lenalidomide will be administered orally with a starting dose of 20mg. Rituximab will be administered intravenously at the standard dose of 375mg/m2. The study will use a standard 3 + 3 design for determination of MTD during cycle 1. There will be three dose levels for escalation, followed by two expansion cohorts of 12 patients each at the MTD, one cohort with follicular lymphoma and one cohort with non-follicular low-grade lymphoma (SLL, marginal zone, lymphoplasmacytic). Patients will be treated for 12 cycles of 4 week duration.
Period: Overall Study
Arm/Group | DL1 (Ixazomib 2.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL2 (Ixazomib 3.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL3/MTD (Ixazomib 4.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | Expansion Cohort I: Follicular Lymphoma at MTD | Expansion Cohort 2: Non-Follicular Lymphoma at MTD
Started | 3 | 3 | 6 | 7 | 0
Completed | 2 | 2 | 1 | 6 | 0
Not Completed | 1 | 1 | 5 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Transformation before study began | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants enrolled in study
Groups:
- Expansion Cohort 1: Follicular Lymphoma at MTD; Expansion Cohort 2: Non-Follicular Lymphoma at MTD: Ixazomib will be orally administered with a starting dose of 2.0mg. Lenalidomide will be administered orally with a starting dose of 20mg. Rituximab will be administered intravenously at the standard dose of 375mg/m2. The study will use a standard 3 + 3 design for determination of MTD during cycle 1. There will be three dose levels for escalation, followed by two expansion cohorts of 12 patients each at the MTD, one cohort with follicular lymphoma and one cohort with non-follicular low-grade lymphoma (SLL, marginal zone, lymphoplasmacytic). Patients will be treated for 12 cycles of 4 week duration.
- Total: Total of all reporting groups
Arm/Group | DL1 (Ixazomib 2.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL2 (Ixazomib 3.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL3/MTD (Ixazomib 4.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | Expansion Cohort 1: Follicular Lymphoma at MTD | Expansion Cohort 2: Non-Follicular Lymphoma at MTD | Total
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 0 | 19
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 0 | 0 | 1 | 1 | 0 | 2
  50-59 years | 2 | 2 | 2 | 1 | 0 | 7
  60-69 years | 0 | 0 | 1 | 4 | 0 | 5
  70-79 years | 1 | 1 | 2 | 0 | 0 | 4
  80-89 years | 0 | 0 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 4 | 0 | 10
  Male | 1 | 2 | 3 | 3 | 0 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6 | 7 | 0 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1
  White | 2 | 3 | 6 | 7 | 0 | 18
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 7 |  | 19

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Oral Ixazomib
Description: To determine the MTD of the combination of oral ixazomib and lenalidomide plus rituximab in patients with previously untreated low-grade B cell lymphoma having high tumor burden by GELF criteria or FLIPI 3-5.
  MTD will be determined using the first 12 participants 15 months after beginning treatment
Time Frame: 15 months after beginning treatment
Population: First 12 participants put on study
Measure: Number; unit: mg
Arm/Group | Lenalidomide + Ixazomib + Rituximab
Number analyzed (Participants) | 12
mg | 4

2. Secondary Outcome: Overall Response Rate
Description: These criteria are based on the Revised Response Criteria for Malignant Lymphoma and include the following categories: Complete Response (CR)(Complete disappearance of all detectable clinical evidence of disease, and disease-related symptoms if present prior to therapy), Partial Response (PR) (A ≥ 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or extranodal masses), Stable Disease (SD) (Failing to attain the criteria needed for a PR or CR, but not fulfilling those for progressive disease), Relapse and Progression (PD) (For determination of relapsed and progressive disease, lymph nodes should be considered abnormal if the long axis is more than 1.5 cm, regardless of the short axis).
Time Frame: Up to 15 months after beginning treatment
Population: Participants who received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | DL1 (Ixazomib 2.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL2 (Ixazomib 3.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL3/MTD (Ixazomib 4.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | Expansion Cohort I: Follicular Lymphoma at MTD | Expansion Cohort 2: Non-Follicular Lymphoma at MTD
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 0
Participants
  Complete response | 1 | 2 | 2 | 5 | 0
  Stable Disease | 2 | 0 | 3 | 0 | 0
  Partial Response | 0 | 0 | 1 | 0 | 0
  Relapse and Progression | 0 | 1 | 1 | 0 | 0

3. Secondary Outcome: Duration of Response
Description: Duration of overall response: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
  The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented.
Time Frame: Up to 15 months after beginning treatment
Population: Participants who received treatment
Measure: Median (Full Range); unit: months
Arm/Group | DL1 (Ixazomib 2.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL2 (Ixazomib 3.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL3/MTD (Ixazomib 4.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | Expansion Cohort I: Follicular Lymphoma at MTD | Expansion Cohort 2: Non-Follicular Lymphoma at MTD
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 0
months | 2.7 [2.7 to 2.7] | 8.9 [2.7 to 15.0] | 5.5 [2.7 to 12.2] | 8.7 [2.8 to 12.9] |

4. Secondary Outcome: Time to Progression
Description: Duration of time from start of treatment to time of progression.
Time Frame: Up to 15 months after beginning treatment
Population: Participants who received treatment
Measure: Median (Full Range); unit: months
Arm/Group | DL1 (Ixazomib 2.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL2 (Ixazomib 3.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL3/MTD (Ixazomib 4.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | Expansion Cohort I: Follicular Lymphoma at MTD | Expansion Cohort 2: Non-Follicular Lymphoma at MTD
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 0
months | 0 [0 to 0] | 2.5 [2.5 to 2.5] | 9.0 [9.0 to 9.0] | 4.6 [4.6 to 4.6] |

5. Secondary Outcome: Progression Free Survival
Description: A number of participants who survived without disease progression
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 15 months after beginning treatment
Population: Participants who received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | DL1 (Ixazomib 2.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL2 (Ixazomib 3.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL3/MTD (Ixazomib 4.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | Expansion Cohort I: Follicular Lymphoma at MTD | Expansion Cohort 2: Non-Follicular Lymphoma at MTD
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 0
Participants | 3 | 2 | 5 | 5 | 0

6. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure (event-free survival) is defined as the time from study entry to first event of disease progression, discontinuation of treatment for any reason, initiation of new treatment, or death.
Time Frame: Up to 15 months after beginning treatment
Population: Participants who received treatment
Measure: Median (Full Range); unit: months
Arm/Group | DL1 (Ixazomib 2.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL2 (Ixazomib 3.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL3/MTD (Ixazomib 4.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | Expansion Cohort I: Follicular Lymphoma at MTD | Expansion Cohort 2: Non-Follicular Lymphoma at MTD
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 0
months | 10 [10 to 10] | 0 [0 to 0] | 6.1 [2.7 to 14.5] | 5.8 [5.8 to 5.8] |

7. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the date of study entry to the date of death.
Time Frame: Up to 15 months after beginning treatment
Population: Participants who received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | DL1 (Ixazomib 2.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL2 (Ixazomib 3.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL3/MTD (Ixazomib 4.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | Expansion Cohort I: Follicular Lymphoma at MTD | Expansion Cohort 2: Non-Follicular Lymphoma at MTD
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 0
Participants | 3 | 3 | 6 | 5 | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: 1 participant in arm "Expansion Cohort I: Follicular Lymphoma at MTD" was taken off study before treatment because of transofrmation and was therefore not followed for adverse events
Arm/Group | DL1 (Ixazomib 2.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL2 (Ixazomib 3.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | DL3/MTD (Ixazomib 4.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) | Expansion Cohort I: Follicular Lymphoma at MTD | Expansion Cohort 2: Non-Follicular Lymphoma at MTD
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 1/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/6 | 3/6 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 6/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DL1 (Ixazomib 2.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) (N=3) | DL2 (Ixazomib 3.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) (N=3) | DL3/MTD (Ixazomib 4.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) (N=6) | Expansion Cohort I: Follicular Lymphoma at MTD (N=6) | Expansion Cohort 2: Non-Follicular Lymphoma at MTD (N=0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | NA
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | NA
Lung Infection- Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | NA
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | NA
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0 | NA
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | NA
Acute renal insufficiency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | NA
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | NA
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0 | NA
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DL1 (Ixazomib 2.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) (N=3) | DL2 (Ixazomib 3.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) (N=3) | DL3/MTD (Ixazomib 4.0 mg + Lenalidomide 20 mg + Rituximab 375mg/m2) (N=6) | Expansion Cohort I: Follicular Lymphoma at MTD (N=6) | Expansion Cohort 2: Non-Follicular Lymphoma at MTD (N=0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 5 | NA
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | NA
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | NA
Indeterminate skin eruptions (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | NA
Itchy scalp (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | NA
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 5 | 5 | NA
Bloating (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | NA
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 5 | NA
Abdominal Cramping (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | NA
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | NA
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 4 | NA
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | NA
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | NA
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | NA
Fatigue (General disorders) | 2 | 0 | 2 | 2 | NA
Fever (General disorders) | 0 | 0 | 0 | 1 | NA
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | NA
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | NA
Flu like symptoms (General disorders) | 0 | 1 | 0 | 1 | NA
Chills (General disorders) | 0 | 0 | 1 | 0 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | NA
Upper Respiratory Infection (Infections and infestations) | 2 | 2 | 2 | 0 | NA
Pleuritic Pain (Infections and infestations) | 1 | 0 | 0 | 0 | NA
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0 | NA
Alkaline phosphatase increased (Infections and infestations) | 0 | 0 | 1 | 0 | NA
Alanine aminotransferase increased (Infections and infestations) | 0 | 0 | 1 | 1 | NA
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | NA
MRSA skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | NA
Legionella pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | NA
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | NA
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0 | NA
Superficial Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | NA
Edema (Vascular disorders) | 1 | 1 | 0 | 3 | NA
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | NA
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | NA
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 0 | 1 | NA
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | NA
Radiculitis (Nervous system disorders) | 1 | 0 | 0 | 0 | NA
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 2 | NA
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | NA
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | NA
Petechiae (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | NA
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | NA
Neutrophil count decreased (Investigations) | 1 | 1 | 3 | 2 | NA
Hypernatremia (Investigations) | 0 | 0 | 1 | 0 | NA
Hypokalemia (Investigations) | 0 | 0 | 2 | 0 | NA
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | NA
Platelet count decreased (Investigations) | 1 | 0 | 1 | 2 | NA
Creatinine increased (Investigations) | 0 | 0 | 2 | 2 | NA
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | NA
Knee pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | NA
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | NA
Upper arm pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | NA
Wrist pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | NA
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | NA
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | NA
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | NA
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | NA
Chest pain- cardiac (Cardiac disorders) | 0 | 0 | 0 | 1 | NA
Conduction disorder (Cardiac disorders) | 0 | 0 | 0 | 1 | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | NA
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | NA
Blurred vision (Eye disorders) | 1 | 0 | 0 | 2 | NA
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT02898259/Prot_SAP_002.pdf
  • Informed Consent Form (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT02898259/ICF_001.pdf